CLINICAL TRIAL: NCT01188122
Title: Optimal Endotracheal Cuff Pressure During Hospitalization in Intensive Care Units Using AnapnoGuard 100 System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospitech Respiration (Industry)
Responsible Party: Study Director, Hospitech Respiration
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HST -AG -01
Record Dates: First submitted 2010-08-23; First posted 2010-08-25 (Estimated); Last update posted 2010-08-25 (Estimated); Status verified 2010-08

CONDITIONS: Ventilator Associated Pneumonia
Keywords: VAP
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AnapnoGuard (Experimental)
  Interventions: Device: AnapnoGuard 100

INTERVENTIONS:
Device: AnapnoGuard 100 — Respiratory guard system during mechanical ventilation

SUMMARY:
Hospitech Respiration Ltd has developed the AnapnoGuard system, an innovative system intended to enhance optimal endotracheal tube (ETT) cuff inflation, by monitoring carbon dioxide (CO2) in upper airways of mechanically ventilated patients. Optimal ETT cuff inflation will lead to a reduction of complication rate related to mechanical ventilation procedure.

This study was design in order to evaluate the feasibility of using the AnapnoGuard system.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 (men and woman);
* Patient is admitted to ICU and expected to receive mechanical ventilation for at least 48 hours;
* Normal chest X-ray;
* Connection of the ETT to the AnapnoGuard system less than 6 hours from intubation initiation;
* Signed informed consent by subject's legally acceptable representative.

Exclusion Criteria:

* Patients who had been treated with mechanical ventilation during the last year;
* Fever from known chest/lung origin;
* Patients with facial, oropharyngeal or neck trauma;
* BMI>35;
* Height < 1.6 m;
* Any chest X-ray pathology during the first 24 hours post intubation;
* More than 7 days hospitalization prior to the intubation. Chest/lung infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-04; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Recording the changes in optimal ETT cuff pressure and their effectors during the course of mechanical ventilation and intubation in Intensive Care Unit (ICU). | during intubation (2-14 days)

SECONDARY OUTCOMES:
Adverse events occurrence | During intubation (2-14 days)

CONTACTS AND LOCATIONS:
Overall Officials: Marian Popescu, Dr., Principal Investigator — Spitalu Universitar De Urgenta Elias Hospital
Locations (1):
- Spitalu Universitar De Urgente Elias Hospital, Bucharest, Romania